CLINICAL TRIAL: NCT03932396
Title: A Novel Hepatitis c micrOelimination Program in Non imprisonEd SenTenced With Alternative Measures
Acronym: HONEST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: HONEST
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Hepatotropic Virus Infection; Addictive Behaviours o Conducts; Mental Disease; People Sentenced to Non-custodial Sentences
Keywords: hepatitis C virus; non-custodial sentences; addictive behaviours; Mental disease; Navigator; screening; POCT
MeSH Terms: conditions — Mental Disorders; Hepatitis C | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group of subjects who fulfill the inclusion criteria: All the population condemned to a non-custodial sentence that is presented in the Service of Management of Penalties and Alternative Measures of the Center of Social Insertion (CIS) José Hierro CP Dueso during the study period (March 2019 and March 2021) , with ages between 18 and 79 years (approximately 1000 people / year) and willing to participate (signs the IC).
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention is planned outside of usual clinical practice. Only active screening for hepatotropic virus infection, mainly hepatitis C virus, HIV, and mental illness will be carried out. If any disease is detected, patients will be referred to the corresponding specialized care following the usual clinical practice.

SUMMARY:
The objective of this study is to carry out a Micro-elimination program for HCV infection in a vulnerable population (people sentenced to non-custodial sentences). This group shares certain peculiarities with the prison population (vulnerability, addictions, mental disorders, etc.), is three times higher than the imprisoned population, and is regularly attended by Social Insertion Centers (CIS) in Spain. An additional objective is to link these people with the specific plans of the Government of Cantabria (Chronicity Plan, Care for Serious Mental Disorders, Harm Reduction Programs and the Center for Attention to Drug Addicts) as well as the Extended Bridge Program for Penitentiary Institutions, implementing the figure of a Navigator (a specialized professional in charge of helping subjects overcome barriers). It is an observational study based on the screening of disease in accordance with the recommendations of the health authorities. Once detected, patients will be referred to the corresponding specialized care following the usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* the entire population served in the Management of Penalties and Alternative Measures Service (SGPMA) of the José Hierro SIC, including new admissions within the study period.

Exclusion Criteria:

* they are not willing to participate and do not sign informed consent.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the population condemned to a non-custodial sentence that is presented in the Service of Management of Penalties and Alternative Measures of the Center of Social Insertion (SIC) José Hierro CP Dueso during the study period (March 2019 and March 2021) , with ages between 18 and 79 years (approximately 1000 people / year) and willing to participate (signs the IC).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-10 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects screened for anti-HCV | From march of 2019 to march of 2021
Percentage of anti-HCV positive | From march of 2019 to march of 2021
Number of anti-HCV positive subjects with detectable viremia | From march of 2019 to march of 2021
Percentage of subjects with detectable viremia | From march of 2019 to march of 2021
To detect other comorbidities such as mental disorders, drug dependencies in this population and link these patients with specific health care programs of Penitentiary Institutions (Extended Bridge Program) and the Government of Cantabria (Chronicity and | From march of 2019 to march of 2021
Number of subjects screened for mental illness. | From march of 2019 to march of 2021
Percentage of subjects with mental illness | From march of 2019 to march of 2021
Number of subjects screened for drug addiction | From march of 2019 to march of 2021
Percentage of subjects with drug addiction | From march of 2019 to march of 2021
Number of subjects linked to the Chronicity Program of the Government of Cantabria | From march of 2019 to march of 2021
Percentage of subjects linked to the Chronicity Program of the Government of Cantabria | From march of 2019 to march of 2021
Number of subjects linked to the Extended Bridge program of Penitentiary Institutions | From march of 2019 to march of 2021
Percentage of subjects linked to the Extended Bridge program of Penitentiary Institutions | From march of 2019 to march of 2021
Number of subjects served by the Navigator | From march of 2019 to march of 2021
Number of subjects with an average rating greater than 4 on a Likert scale of 5 points of satisfaction with the Navigator | From march of 2019 to march of 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

REFERENCES:
- [Background] Cuadrado A, Llerena S, Cobo C, Pallas JR, Mateo M, Cabezas J, Fortea JI, Alvarez S, Pellon R, Crespo J, Echevarria S, Ayesa R, Setien E, Lopez-Hoyos M, Crespo-Facorro B, Aguero J, Chueca N, Garcia F, Calleja JL, Crespo J. Microenvironment Eradication of Hepatitis C: A Novel Treatment Paradigm. Am J Gastroenterol. 2018 Nov;113(11):1639-1648. doi: 10.1038/s41395-018-0157-x. Epub 2018 Jun 27. PMID 29946175
- [Result] Blachier M, Leleu H, Peck-Radosavljevic M, Valla DC, Roudot-Thoraval F. The burden of liver disease in Europe: a review of available epidemiological data. J Hepatol. 2013 Mar;58(3):593-608. doi: 10.1016/j.jhep.2012.12.005. PMID 23419824